CLINICAL TRIAL: NCT04943133
Title: Study of the Agreement Between Two Methods of Measuring Brachial Systolic Pressure (SFATI or Auscultatory) in Pregnant Women With or Without Blood Pressure Disorders and Search for Markers of Arterial Stiffness in Pre-eclampsia.
Brief Title: Concordance Between the Systolic Foot-to-Apex Interval and the Auscultatory Method for Measuring Brachial Systolic Pressure in Pregnant Women With or Without Blood Pressure Disorders and Search for Markers of Arterial Stiffness in Pre-eclampsia.
Acronym: SFATI GROPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDIL/2020/APM-001
Record Dates: First submitted 2021-03-15; First posted 2021-06-29 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Blood Pressure Disorders; Pregnancy Induced Hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Blood Pressure Determination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3rd-term group: Pregnant women included in the last 3 months of pregnancy (Active Comparator): Comparison of the profile of the curve according to whether there is presence or absence of blood pressure disorders.
  Interventions: Device: Blood pressure measurement and collection of the oscillometric curve for later SFATI analysis; Device: Blood pressure measurement with the usual equipment used in the department; Device: systematic measurement of pulse wave velocity (aortic and brachial)
- Before 20 weeks group. Pregnant women (normal blood pressure) included before 20 weeks of pregnancy. (Active Comparator): Comparison of the profile of the curve according to the presence or absence of risk factors for pre-eclampsia
  Interventions: Device: Blood pressure measurement and collection of the oscillometric curve for later SFATI analysis; Device: Blood pressure measurement with the usual equipment used in the department

INTERVENTIONS:
Device: Blood pressure measurement and collection of the oscillometric curve for later SFATI analysis — Brachial systolic arterial blood pressure will be systematically taken with acquisition of the oscillometric curve for analysis and measurement with the SFATI system and simultaneous electronic recording of the Korotkoff sound (auscultatory method) and a search for SFATI arterial stiffness markers for all patients. Brachial systolic arterial blood pressure will be measured with the help of a cuff equipped with a Biopac SS30L electronic stethoscope and a MA-300 phonocardiographic microphone, placed side-by-side immediately downstream from the brachial occlusion cuff. The various signals (pneumatic cuff, oscillometric signal and Korotkoff sounds) will be digitalized by an MP35 system.
Device: Blood pressure measurement with the usual equipment used in the department — Brachial systolic blood pressure will be taken via the conventional oscillometric method, only for hospitalized women. Blood pressure will be measured on the same arm with the help of a conventional Dinamap-type automat (GE), with at least 2 minutes between the end of the first measurement and the start of the second inflation.
Device: systematic measurement of pulse wave velocity (aortic and brachial) — Carotid to femoral and carotid to radial pulse wave velocity (Complior) will be systematically determined for hospitalized women and offered to all women seen for consultation.
  Pulse wave velocity will be measured with the help of a Complior tonometric system (Alam Medical, Vincennes, France), with which the aorta and the arterial axes of the upper limb used to measure blood pressure can also be measured.
  Arms: 3rd-term group: Pregnant women included in the last 3 months of pregnancy

SUMMARY:
The investigators hypothesize that the Systolic Foot-to-Apex Time Interval (SFATI) method is an accurate means of measuring systolic blood pressure in pregnant women at a risk of pre-eclampsia. As the presence of arterial calcifications only changes the concordance between the SFATI method and the auscultatory reference method if calcifications are very severe, it should make it possible to identify, at an early stage, those women with a higher risk of developing pre-eclampsia. This is a transversal study with monocentric prospective recruitment to evaluate a non-CE (Conformité Européenne) -marked medical device in a diagnostic situation.

DETAILED DESCRIPTION:
During pregnancy, high blood pressure remains the leading cause of maternal and foetal morbidity and mortality due to its complications and affects 5 to 10% of pregnancies. Hypertension in pregnancy is based on measurements taken in a medical setting and is defined by a systolic blood pressure ≥ 140 mmHg and/or a diastolic ≥ 90 mmHg. Regular monitoring of blood pressure is therefore recommended during pregnancy.

However, the main difficulty lies in the unreliability of many measuring devices. One of the hypotheses that may explain this unreliability is that they are based on the analysis of the oscillometric curve. The latter is influenced by the behaviour of the arterial wall and its biomechanical properties. However, during normal pregnancy, arterial compliance is altered, particularly as a result of hypervolaemia. With hypertension and pre-eclampsia, these changes are even more pronounced.

The gold standard for measuring blood pressure remains the auscultatory method based on the detection of Korotkoff's sounds. Now, this method is being used less and less in favour of the oscillometric method and increasing use of automated devices.However, these automatons use algorithms that are neither revealed nor interchangeable and, despite them being CE marked, the majority of the devices on the market have not been validated by clinical trials in accordance with the recommendations. Validating them in pregnant women is even more problematic and it is generally accepted that most voltage measurement systems can be faulty. To improve the accuracy and reproducibility of the oscillometric method, we have developed a new algorithm for determining systolic blood pressure based on the oscillometric curve, involving a temporal analysis of the oscillometric curve, not its envelope. This original approach has made it possible to highlight an increase in the delay between the foot and the peak of the systolic peak of the oscillogram (SFATI - Systolic Foot-to-Apex Time Interval), the maximum value of which coincides with the first Korotkoff sound, thus allowing real measurement of systolic blood pressure for the first time, not just a calculation.

In addition, this parameter presents a second elevation, observed in the region of mean blood pressure in patients with cardiovascular risk factors and therefore at a risk of increased arterial stiffness. This parameter should make it possible to easily identify subjects with an arterial compliance disorder via a simple standard blood pressure measurement. This opens up many possibilities in terms of screening including on a large scale and repeated basis.

Thus, with a simple blood pressure measurement, the SFATI algorithm should make it possible to correct the inconsistencies observed with the conventional oscillometric method during pregnancy, with two advantages :

* precise, reliable blood pressure measurement ensuring not only the diagnosis of pre-eclampsia but also the quality of monitoring, which is a prerequisite for appropriate therapeutic management;
* evaluation of the vessel walls, by detecting possible stiffness, indicating arterial damage. The aim here is to characterise the curve profile obtained in women with pre-eclampsia, at various levels of severity and also to evaluate this profile in women with a history of pre-eclampsia or at risk of pre-eclampsia. The possible specificities would then make it possible to integrate this approach into the current screening strategy in order to evaluate its interest on a larger scale.

We therefore make the following assumptions :

1. the SFATI method is more reliable than the standard auscultatory method for accurately measuring brachial systolic blood pressure in pregnant women, whatever their blood pressure status;
2. in women with blood pressure disorders, the oscillometric curve is modified with the presence of arterial stiffness markers, making it possible to characterise a particular oscillometric profile.
3. this particular profile appears at an early stage and should make it possible to identify women at higher risk of developing pre-eclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Patient monitored for a single pregnancy in consultation or hospitalized in the department of Gynecology-Obstetrics at Nîmes University Hospital.
* Patient has given written informed consent.
* Patient has signed the consent form.
* Patient is covered by a health insurance scheme.
* Patient is aged over 18.

Exclusion Criteria:

* Multiple pregnancy.
* Patient is taking part in a category 1 research study.
* Patient is in a period of exclusion determined by another study.
* Patient is under legal protection or curatorship.
* Patient is in no condition to express her consent.
* Patient for whom it is impossible to give clear information.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 132 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure in pregnant women whatever the gestational age : Auscultatory method | Inclusion visit, Day 0
  The brachial systolic blood pressure of pregnant women with or without hypertensive disorders will be measured by the standard auscultatory method based on the Korotkoff sounds, in mmHg.
Systolic blood pressure in pregnant women whatever the gestational age : SFATI method. | Inclusion visit, Day 0
  The brachial systolic blood pressure of pregnant women with or without hypertensive disorders will be measured by the SFATI (Systolic Foot-to-Apex Time Interval) method.
Concordance between the auscultatory method and the SFATI method for measuring systolic blood pressure in pregnant women whatever the gestational age. | Inclusion visit, Day 0
  Lin's concordance correlation coefficient will be used to compare the simultaneous recording of Korotkoff sound and the brachial systolic pressure using the SFATI method. Good if the lower limit of the 95% confidence interval is >0.9 and ACCEPTABLE if the lower limit is >0.8.
Presence or not of hypertensive disorders revealed using the SFATI method. | Inclusion visit, Day 0
  YES/NO
Type of hypertensive disorders. | Inclusion visit, Day 0.
  If hypertensive disorders are revealed, these will be described along with the gestational age at which they were discovered.

SECONDARY OUTCOMES:
Systolic blood pressure in pregnant women whatever the gestational age : Oscillatory method (Dinamap). | Inclusion visit, Day 0
  The brachial systolic blood pressure of pregnant women with or without hypertensive disorders will be measured by the standard oscillatory method (Dinamap) in mmHg.
Concordance between the SFATI method and the conventional oscillatory method for blood pressure monitoring (Dinamap), in pregnant women with or without hypertensive disorders, whatever the gestational age. | Inclusion visit, Day 0
  Lin's concordance correlation coefficient will be used to compare the brachial systolic pressure obtained with the oscillatory method and using the SFATI method. GOOD if the lower limit of the 95% confidence interval is >0.9 and ACCEPTABLE if the lower limit is >0.8.
Concordance between the conventional oscillatory method (Dinamap), and the auscultatory method for blood pressure monitoring in pregnant women with or without hypertensive disorders, whatever the gestational age. | Inclusion visit, Day 0
  Lin's concordance correlation coefficient will be used to compare the brachial systolic pressure obtained with the oscillatory method and using the auscultatory method. GOOD if the lower limit of the 95% confidence interval is >0.9 and ACCEPTABLE if the lower limit is >0.8.
Profile of the oscillometric curve processed by the SFATI algorithm. Last term of pregnancy in normal pregnancies. | Inclusion visit, Day 0
  Presence of hypertensive disorders.YES/NO.
Profile of the oscillometric curve processed by the SFATI algorithm. Last term of pregnancy in women with hypertensive disorders or pre-eclampsia. | Inclusion visit, Day 0
  Presence of hypertensive disorders.YES/NO.
Profile of the oscillometric curve processed by the SFATI algorithm before 20 weeks of pregnancy in women with or without a risk of hypertensive disorders. | Inclusion visit, Day 0
  Presence of a second peak on the oscillometric curve.YES/NO.
Profile of the oscillometric curve processed by the SFATI algorithm according to aortic pulse wave velocity in women with (>9 m/s) or with no acceleration of aortic pulse wave velocity. | Inclusion visit, Day 0
  Presence of a second peak on the oscillometric curve.YES/NO.
Profile of the oscillometric curve processed by the SFATI algorithm according to brachial pulse wave velocity in women with (>12 m/s) or with no acceleration of brachial pulse wave velocity. | Inclusion visit, Day 0
  Presence of a second peak on the oscillometric curve.YES/NO.

CONTACTS AND LOCATIONS:
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France